CLINICAL TRIAL: NCT02274961
Title: S-pantoprazole 10mg Phase III Clinical Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LTP10_KR_1301
Record Dates: First submitted 2014-10-13; First posted 2014-10-27 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Non Erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-pantoprazole 10mg (Experimental): S-pantoprazole 10mg Tablet once daily for 4 weeks
  Interventions: Drug: S-pantoprazole 10mg
- Placebo (Placebo Comparator): Placebo tablet for the test drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-pantoprazole 10mg
  Arms: S-pantoprazole 10mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This clinical study hypothesized that S-pantoprazole 10mg would be effective to treat Non erosive Reflux Disease than placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 19 and 75 inclusive
* Patient with a history of heartburn or acid regurgitation for at least 3 months.
* Those with episodes of heartburn for 2 days or more during the last 7 days prior to baseline
* Patients negative for erosive esophagitis confirmed by esophagogastroduodenoscopy(EGD) performed within 7 days of screening
* Capable of providing written informed consent, willing and able to a comply with all procedures of the study

Exclusion Criteria:

* History of endoscopic erosive esophagitis(EE) at screening EGD.
* Historical evidence of the following disease/conditions : symptom of Irritable bowel syndrome
* More tha 3cm endoscopic Barrett's esophagus or significant dysplastic changes in the esophagus
* Proton Pump Inhibitor(PPI) within 4 weeks prior to the baseline visit
* H2-receptor antagonist, sucralfate, prokinetics, Non Steroidal Antiinflammatory Drugs(NSAIDs) (except low dose aspirin) during the 2 weeks prior to the screening
* Historical evidence of the following disease/conditions during 3 months: Zollinger-Ellison syndrome, the primary esophageal motility disorders achalasia, esophageal stricture, pancreatitis, gastric ulcer, evidence of upper G.I. malignancy, pancreatitis, malabsorption, severe cardiovascular or pulmonary disease, severe liver disease, severe renal disease, cerebral vascular disease,
* Known hypersensitivity to any component of drug
* pregnancy or lactation (F only)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy , as defined by complete resolution of heartburn (HB) per Questionnaire, of 4 weeks of treatment of S-pantoprazole 10mg qd compared to Placebo in subjects with symptomatic gastro-esophageal reflux disease | 4 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Yeungnam University Medical Center, Daegu, Daegu
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si, Gyeonggi-do
  - Bundang CHA Medical Center, Sung-Nam, Gyeonggi-do
  - Seoul National University Bundang Hospital, Sung-Nam, Gyeonggi-do
  - Asan Medical Center, Seoul, Seoul
  - Gangnam Severance Hospital, Seoul, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, Seoul
  - Seoul National University Hospital, Seoul, Seoul
  - Severance Hospital, Seoul, Seoul
  - Seoul St. Mary's Hospital, Seoul